CLINICAL TRIAL: NCT05416086
Title: iCLAS™ Cryoablation System Post-Market Clinical Follow-up (PMCF) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adagio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-086
Record Dates: First submitted 2022-06-07; First posted 2022-06-13 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCLAS Cryoablation arm (Other): all subjects will receive a cryoablation procedure with the iCLAS System and be followed up for 12-month
  Interventions: Device: cryoablation procedure using the iCLAS Cryoablation System

INTERVENTIONS:
Device: cryoablation procedure using the iCLAS Cryoablation System — all subjects will receive a cryoablation procedure using the iCLAS Cryoablation System (catheter, stylets, and console) and warming balloon

SUMMARY:
A prospective, single-arm, multi-center study designed to collect real world safety and performance data of the Adagio Medical iCLAS Cryoablation System in the treatment of drug refractory, recurrent, symptomatic, Paroxysmal Atrial Fibrillation (PAF), Persistent Atrial Fibrillation (PsAF), and Atrial Flutter (AFL).

DETAILED DESCRIPTION:
This Post-Market Clinical Follow-up (PMCF) study continues collecting additional information about the Adagio Medical iCLAS™ Cryoablation System in real world clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Planned ablation procedure according to the indication for use of the commercially available Adagio iCLAS™ Cryoablation System
* Subject willing to comply with study requirements and give informed consent.

Exclusion Criteria:

* In the opinion of the Investigator, any known contraindication to an atrial ablation procedure with the Adagio iCLAS™ Cryoablation System as indicated in the device Instructions For Use (IFU).
* Subject is enrolled in a study that has not been approved for concurrent enrollment by the sponsor.
* Any other condition that, in the judgment of the investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, terminal illness with a life expectancy of less than one year, extensive travel away from the research center)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome - freedom from AF | 12 months
  Freedom from Atrial Fibrillation (AF) recurrence during the 12-months follow-up period.
Primary outcome - freedom from AF/AT/AFL | 12 months
  Freedom from Atrial Arrhythmia at 12-months
Primary outcome - freedom from Device/Procedure Related Adverse Events | during procedure and up to 12-month follow up
  Freedom from Device / Procedure Related Adverse Events during and after the ablation procedure through12-month follow up

CONTACTS AND LOCATIONS:
Locations (4):
- Onze-Lieve-Vrouw Hospital Aalst (OLV), Aalst, Belgium
- Universitatsklinikum Erlangen, Erlangen, Germany
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No